CLINICAL TRIAL: NCT00162630
Title: Fascia Iliaca Compartment Blockade as Analgesia for Hip Fractures in the Acute Phase
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: IMK Fonden (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: HHSG-rct-04
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2006-09-15 (Estimated); Status verified 2006-09

CONDITIONS: Hip Fracture
Keywords: Hip fracture, pain, regional anaesthesia, analgesia
MeSH Terms: conditions — Hip Fractures; Pain; Agnosia

INTERVENTIONS:
Procedure: Fascia Iliaca Compartment Blockade

SUMMARY:
To evaluate the analgesic potential of an neural blockade (Fascia iliaca compartment) with local anaesthetics in patients with hip fracture immediately after arrival in the emergency department.

DETAILED DESCRIPTION:
Hip fracture patients have severe pain in the acute phase. Traditional analgesic treatment have consisted of intramuscular morphine with its associated side effects. The trial evaluates the Fascia iliaca compartment compared to regular opioid pain therapy in hip fracture patinets immediately after arrival at the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* Primary hip fracture suspected
* able to give informed consent
* no substance abuse
* no regular opioid therapy
* no opioid treatment within the last 6 hours
* morphine intolerance
* allergies to local anaesthetics

Exclusion Criteria:

* Fracture ruled out on x-ray

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2003-05; Study Completion 2006-03

PRIMARY OUTCOMES:
Pain relief within 3 hours

SECONDARY OUTCOMES:
Nausea
Pain on transfer
Discomfort with block placement

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai B Foss, MD, Study Director — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

REFERENCES:
- [Derived] Guay J, Kopp S. Peripheral nerve blocks for hip fractures in adults. Cochrane Database Syst Rev. 2020 Nov 25;11(11):CD001159. doi: 10.1002/14651858.CD001159.pub3. PMID 33238043